CLINICAL TRIAL: NCT06135051
Title: Deep Brain Therapy With Low-intensity Ultrasound for Treatment of Cognitive Impairment
Brief Title: Ultrasonic Neuromodulation for Treatment of Cognitive Impairment
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IRB administrative closure
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jan Kubanek, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00173042
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Dementia; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active stimulation (Experimental): Low-intensity transcranial focused ultrasound stimulation of deep brain targets affected by Alzheimer's disease.
  Interventions: Device: Diadem prototype
- Sham stimulation (Sham Comparator): Sham stimulation that applies the device in the same way as verum but only delivers auditory sounds correspoding to the ultrasonic pulses.
  Interventions: Device: Diadem prototype

INTERVENTIONS:
Device: Diadem prototype — The device delivers low-intensity ultrasonic waves into specific brain targets.

SUMMARY:
This study will evaluate a new form of non-invasive deep brain therapy for individuals with Alzheimer's disease. Low-intensity transcranial focused ultrasound stimulation will first be delivered using a range of stimulation parameters during psychophysical and physiological monitoring. A well-tolerated stimulation protocol will be selected for subsequent testing in a blinded randomized sham-controlled cross-over trial. The trial will evaluate brain target engagement using magnetic resonance imaging, PET imaging, and numerical scales of cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment or mild dementia due to Alzheimer's disase (AD) with confirmed AD biomarkers (Amyloid PET or CSF)
* Age 65-80
* MOCA > 18

Exclusion Criteria:

* Evidence of cerebral amyloid angiopathy or stroke within 1 year
* Clinical symptoms or findings suggestive of alternative diagnosis or co-pathology
* Inability to complete MRI
* Suicidal ideation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-08-18 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Test for Dementia (MoCA) | Up to 3 months following study initiation
  The MoCA is a 30-point test to detect cognitive impairment. Scores range from 0 (poor) and 30 (perfect).
Hamilton Depression Rating Scale (HDRS-17) | Up to 3 months following study initiation
  This 17-item questionnaire rates the severity of depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. The scores range from 0 (no symptoms) to 52 (worst possible).
Amyloid PET | Up to 3 months following study initiation
  PET (positron emission tomography) combined with fluorine-18 labelled radiotracers provide brain scans that are interpreted as either amyloid-beta positive or negative.

SECONDARY OUTCOMES:
Hopkins Verbal Learning Test-Revised (HVLT-R) | Up to 3 months following study initiation
  HVLT-R is a verbal memory test with 12 words learned over three trials, with the correct words summed for the Total Recall score (range = 0 (worst) - 36 (best)). The Delayed Recall score is the number of correct words recalled after a 20 - 25-minute delay (range = 0 (worst) - 12 (best)).
Digit Span Memory Test | Up to 3 months following study initiation
  A standard test for working memory. In this test, a list of random numbers or letters is presented on a computer screen at the rate of one per second. The test begins with three numbers, increasing until the person commits errors. The average digit span for normal adults without error is seven plus or minus two. The higher the number, the more patent the working memory.
Trail Making Test, Part A and B | Up to 3 months following study initiation
  The test probes visual scanning and working memory. The task is to connect a set of 25 dots as quickly as possible while maintaining accuracy. The faster the completion of Part A and Part B, the better.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No